CLINICAL TRIAL: NCT01880450
Title: Longitudinal Intervention Study to Prepare Early Adolescents for Middle Adolescence, Specifically Focusing on Improving Sexual Health Outcomes
Brief Title: Project Prepared: Risks, Roles and Relationships
Acronym: Prepared
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Laurie Bauman, Professor; Director, Preventive Intervention Research Center, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2008-551; 5R01HD062079 (NIH)
Record Dates: First submitted 2011-07-12; First posted 2013-06-19 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: F01.145.802.845; F01.145.802.987

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Project Prepared (Experimental)
  Interventions: Behavioral: Project Prepared
- TEEN-Teen Education & Employment Network (Active Comparator)
  Interventions: Behavioral: TEEN

INTERVENTIONS:
Behavioral: Project Prepared — Behavioral intervention to reduce sexual risk and promote healthy relationships
  Arms: Project Prepared
Behavioral: TEEN — Control condition the promote communication, decision-making skills etc.
  Arms: TEEN-Teen Education & Employment Network

SUMMARY:
Project Prepared is a theoretically based, comprehensive, intensive group intervention that is designed to prepare early adolescents for middle adolescence and its challenges. It emphasizes skills in avoiding risky sexual situations, and provides medically accurate information about sexual development, sexually transmitted infections and pregnancy. Effectiveness is measured by using a randomized control trial design and tracking differences in cognitive factors (HIV/STI (Sexually Transmitted Infections) knowledge, sexual self-efficacy; intention to use a condom); relationship factors (immature romantic beliefs, relationship self-efficacy), gender norms (macho man, powerless female), and resilience.

ELIGIBILITY:
Inclusion Criteria:

* 12-14 yrs old
* lives in the Bronx, NY at Baseline
* Has been seen at some point in one of the Montefiore Medical Center community health clinics.

Exclusion Criteria:

* Inability to independently complete the questionnaire/training due to sensory, cognitive or motor disabilities.
* Reading ability NOT at 5th grade on the reading subtest of the Wide-range Achievement Test.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 397 (Actual)
Dates: Start 2009-05; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Intentions to engage in safer sex behavior at 6 months | 6 months post baseline
  measuring change from baseline to 6 months (as compared to control group)
Change in Intentions to engage in safer sex behavior at 1 year | 1 year post baseline
  measuring change from baseline to 1 year (as compared to control group)

SECONDARY OUTCOMES:
Change in Cognitive Factors at 6 months | 6 months post baseline
  measuring change in HIV/STI knowledge, condom outcome and efficacy expectancies, sexual self-efficacy from baseline to 6 months (compared to control group)
Change in Cognitive Factors at 1 year | 1 year post baseline
  measuring changes in HIV/STI knowledge, condom outcome and efficacy expectancies, sexual self-efficacy from baseline to 1 year (as compared to control group)

CONTACTS AND LOCATIONS:
Overall Officials: Laurie J Bauman, PhD, Principal Investigator — Albert Einstein College of Medicine, Pediatrics Division
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

REFERENCES:
- [Derived] Bauman LJ, Watnick D, Silver EJ, Rivera A, Sclafane JH, Rodgers CRR, Leu CS. Reducing HIV/STI Risk Among Adolescents Aged 12 to 14 Years: a Randomized Controlled Trial of Project Prepared. Prev Sci. 2021 Nov;22(8):1023-1035. doi: 10.1007/s11121-021-01203-0. Epub 2021 Feb 19. PMID 33606173